CLINICAL TRIAL: NCT02480335
Title: The Clinical Efficacy And Subclinical Effects on Arterial STIFFNESS of Bosentan Therapy Added to Usual Care in Patients With Systemic Sclerosis With Digital Ulcers
Brief Title: The Clinical And Subclinical Effects on Arterial Stiffness of Bosentan in Patients With Systemic Sclerosis
Acronym: CEASESTIFF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, dr. DJ Mulder, dr. Douwe J. Mulder, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL49919.042.14
Record Dates: First submitted 2015-06-15; First posted 2015-06-24 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care and bosentan (Experimental): Usual care and also treatment with bosentan.
  Interventions: Drug: bosentan
- Usual care (No Intervention): Usual care only.

INTERVENTIONS:
Drug: bosentan — 62.5 mg oral twice daily for 4 weeks, then 125 mg oral twice daily.
  Other Names: tracleer
  Arms: Usual care and bosentan

SUMMARY:
The aim of the study is to investigate whether bosentan added to usual care improves arterial stiffness after 3 months as measured as the pulse wave velocity (PWV) of the medium and large arteries corrected for blood pressure changes in patients with systemic sclerosis (SSc) with digital ulcers (DU). Patients will be randomized into a group with usual care and bosentan (n=10) or usual care only (n=10). PWV will be assessed at baseline, 3 months and 12 months.

DETAILED DESCRIPTION:
Rationale: Digital ischemia is a major problem in patients with Raynaud's phenomenon (RP), especially in those with underlying connective tissue diseases such as systemic sclerosis (SSc). SSc is hallmarked by microvascular disease which can be assessed by nailfold capillary microscopy (NCM) to identify specific capillary patterns. However, it appears that vascular damage is not restricted to the capillaries, but may also extend to more upstream hand and forearm arteries. This may not only be reflected by clinically relevant structural abnormalities such as obliteration, but also by decreases in arterial function. The best characterised in RP is the occurrence of vasospasms after cold exposure. However, evidence points out that major stiffening of the arteries also occurs, potentially exaggerating digital ischemia and other vascular complications in SSc.

Objective: To investigate whether bosentan added to usual care improves arterial stiffness after 3 months as measured as the pulse wave velocity of the medium and large arteries corrected for blood pressure changes in patients with systemic sclerosis with digital ulcers.

Intervention:

Group 1: Usual care AND bosentan 62.5 mg twice daily, titrated to 125 mg twice daily after one month if tolerated (n=10) Group 2: Usual care only (n=10)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Bosentan is a registered product in the Netherlands. In this study, it will be used within its indication and not in combination with other products for which it has not been registered. Therefore no additional unknown uncertainties and increased overall risk are applicable for the investigational product. In the usual care group, treatment will not differ from clinical practice. To minimize the risk of patients not receiving the most appropriate treatment in the control group, regular visits and lab assessments are planned. Patients are allowed to start with bosentan in the usual care group if indicated by the treating physician. The study will consist of one screening and three study visits. During the latter, patients clinical signs and symptoms will be assessed, vascular lab will be performed, blood will be drawn, and subjects be asked to fill in questionnaire, all of which will have a duration of no more than 2 hours per visits. In total 3 times 24cc of blood will be collected, preferably in combination will routine lab assessments. These measures render the risks acceptable and the burden minimal for the subjects participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Systemic sclerosis based on the 2013 American College of Rheumatology/European League Against Rheumatism criteria
* Raynaud's phenomenon
* A history of digital ulcer disease
* Assessable Pulse Wave Velocity measurement at baseline
* Written informed consent

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Systolic blood pressure lower than 85 mmHg
* Moderate to severe hepatic impairment, i.e., Child-Pugh class B or C
* Baseline values of liver aminotransferases, i.e., aspartate aminotransferases and/or alanine aminotransferases, greater than 3 times the upper limit of normal
* Concomitant use of cyclosporine A
* Pregnancy
* Women of child-bearing potential who are not using reliable methods of contraception
* Significant peripheral vascular disease as the sole consequence of atherosclerotic disease due to conventional vascular risk factors and coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Mean of right and left carotid-femoral arterial (i.e. aortic) Pulse Wave Velocity (cfPWV) | 3 months
  assessed with Sphygmocor

SECONDARY OUTCOMES:
Mean of right and left carotid-femoral arterial (i.e. aortic) Pulse Wave Velocity (cfPWV) | 12 months
  assessed with Sphygmocor
Right carotid-brachial arterial PWV (cbPWV) | 3 and 12 months
  assessed with Sphygmocor
Left carotid-brachial arterial PWV (cbPWV) | 3 and 12 months
  assessed with Sphygmocor
Right carotid-radial arterial PWV (crPWV) | 3 and 12 months
  assessed with Sphygmocor
Left carotid-radial arterial PWV (crPWV) | 3 and 12 months
  assessed with Sphygmocor
Local PWV of the right radial artery (rPWV) | 3 and 12 months
  ultrasound assessment using a MyLabOne Vascular machine
Local PWV of the left radial artery (rPWV) | 3 and 12 months
  an ultrasound assessment using a MyLabOne Vascular machine
Local PWV of the right brachial artery (bPWV) | 3 and 12 months
  an ultrasound assessment using a MyLabOne Vascular machine
Local PWV of the left brachial artery (bPWV) | 3 and 12 months
  an ultrasound assessment using a MyLabOne Vascular machine
Microangiopathy Evolution Score (MES) | 3 and 12 months
  With nailfold capillary microscopy
Capillaroscopic Skin Ulcer Risk Index (CSURI) | 3 and 12 months
  With nailfold capillary microscopy
Prognostic Index for Digital Lesions (PILD) | 3 and 12 months
  With nailfold capillary microscopy
Mean widened capillaries of 8 fingers (dig 2-5) | 3 and 12 months
  number per finger, assessed with nailfold capillary microscopy
Mean giant capillaries of 8 fingers (dig 2-5) | 3 and 12 months
  number per finger, assessed with nailfold capillary microscopy
Mean capillary density of 8 fingers (dig 2-5) | 3 and 12 months
  number per mm per finger, assessed with nailfold capillary microscopy
Mean loop width of 8 fingers (dig 2-5) | 3 and 12 months
  mm per capillary per finger, assessed with nailfold capillary microscopy
Blood flow in the hands in region of interest (ROI) 1: distal of the proximal interphalangeal (PIP) joint of the 3 middle fingers | 3 and 12 months
  Measured by Laser Doppler Perfusion Imaging
Blood flow in the hands in ROI 2: distal of the metacarpal joints and proximal of the PIP joint | 3 and 12 months
  Measured by Laser Doppler Perfusion Imaging
Blood flow in the hands in ROI 3: the hand proximal of the metacarpal joints | 3 and 12 months
  Measured by Laser Doppler Perfusion Imaging
Skin Autofluorescence | 3 and 12 months
  assessed with the AGE Reader
Number of new digital ulcers | 3 and 12 months
  Number
Time to healing of digital ulcers | 3 and 12 months
  In days
Urine albumin/creatinine ratio (ACR) | 3 and 12 months
  Measured in two separate morning samples of urine
Plasma N-terminal of the prohormone brain natriuretic peptide (NT-proBNP) | 3 and 12 months
  assessed using a routine assay
Serum levels of matrix metalloproteinase 3 | 3 and 12 months
  measured according to the manufacturer's instructions
Serum levels of matrix metalloproteinases 9 | 3 and 12 months
  determined using in-house enzyme-linked immunosorbent assays (ELISAs)
Serum levels of tissue inhibitors of metalloproteinases (TIMP) | 3 and 12 months
  determined using in-house enzyme-linked immunosorbent assays
Blood pressure of the brachial artery | 3 and 12 months
  systolic/diastolic in mmHg
Modified Rodnan Skin Score (mRSS) | 3 and 12 months
  17 body areas are examined by clinical palpation and scored based on examiner judgement of skin thickness on a 4-point ordinal scale.
Scleroderma Health Assessment Questionnaire (SHAQ) | 3 and 12 months
  questionnaire
Short Form (36) | 3 and 12 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andries J Smit, MDPhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands